CLINICAL TRIAL: NCT04262180
Title: Multi-site Adaptive Trial of a Technology-based, EHR-integrated Physical Activity Intervention in Breast and Endometrial Cancer Survivors
Brief Title: Physical Activity Promotion for Breast and Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Northwestern University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-1361; EDUC/KINESIOLOGY/KINESIOLOG (Other: UW Madison); 1R37CA225877-01A1 (NIH); A176000 (Other: University of Wisconsin, Madison); UW18094 (Other: UW Madison); Protocol Version 2/22/2024 (Other: UW Madison); NCI-2020-00400 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Physical Activity; Breast Cancer Survivors; Endometrial Cancer Survivors
Keywords: MVPA; Fitbit
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: One control arm and two randomized arms. Every participant starts with a base intervention, non-responders will be randomized to one of the two arms.
Who Masked: Outcomes Assessor
Masking Description: Stratified randomization. Assessors will be blinded to which arm the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Base intervention- Fitbit with EHR integration (Experimental): All participants will receive a first-line intervention (i.e., Fitbit activity tracker with EHR integration including messages delivered via the EHR's patient portal) and will be evaluated for response/non-response every 4 weeks until week 20.
  Interventions: Other: Base intervention-Fitbit with EHR integration
- Nonresponders -Stepped up to Online gym (Experimental): Non-responders to 'fitbit with EHR integration' will be randomized to be "stepped up" to one of two augmentation strategies(either Online gym or coaching calls). This arm will be stepped up to Online gym.
  Interventions: Other: Base intervention-Fitbit with EHR integration; Other: Online Gym
- Nonresponders -Stepped up to Coaching calls (Experimental): Non-responders to 'fitbit with EHR integration' will be randomized to be "stepped up" to one of two augmentation strategies(either Online gym or coaching calls). This arm will be stepped up to Coaching calls.
  Interventions: Other: Base intervention-Fitbit with EHR integration; Other: Coaching Calls

INTERVENTIONS:
Other: Base intervention-Fitbit with EHR integration — Every subject will start with a base intervention - Fitbit activity tracker with EHR integration including messages delivered via the EHR's patient portal
Other: Coaching Calls — Non-responders to base intervention will be randomized to coaching calls.
  Arms: Nonresponders -Stepped up to Coaching calls
Other: Online Gym — Non-responders to base intervention will be randomized to online gym.
  Arms: Nonresponders -Stepped up to Online gym

SUMMARY:
Many breast and endometrial cancer survivors do not get enough physical activity. Technology-based interventions can be inexpensive and easy to scale up, however they are not effective for all women. The purpose of this study is test an adaptive physical activity intervention approach that reserves the most resources and support for women who do not fare well with a lower-cost, minimal intervention. The results from this trial will inform the development of scalable physical activity interventions for breast and endometrial cancer survivors.

DETAILED DESCRIPTION:
There are 3,000,000 breast and 760,000 endometrial cancer survivors in the US and these populations will grow 30% by 2026. Increased moderate-to-vigorous intensity physical activity (MVPA) is consistently associated with enhanced quality of life, reduced chronic disease risk, and improved cancer prognosis in these survivors yet 70-90% fail to engage in the 150 minutes/week of MVPA recommended by the American Cancer Society. Unfortunately, since physical activity support is not a part of standard survivorship care, few survivors have access to efficacious MVPA interventions. A key barrier to translation of MVPA promotion into care is the design of existing programs, which are resource-intensive, costly, and deliver multiple components (i.e., coaching calls, supervised exercise) simultaneously to all participants. This "one-size-fits-all" approach does not account for individual needs, nor can it realistically be implemented into care. Thus there is a critical need for effective, scalable interventions that efficiently allocate resources to meet each woman's needs.

An adaptive approach that tries minimal, low resource treatments (i.e., technology tools) for everyone first, and reserves the use of higher-resource components (e.g., coaching) for survivors who fail to increase MVPA, offers a promising alternative to traditional approaches. This engages women who lack the time or transportation to participate in more intensive interventions, yet avoids providing high-resource components to those who would respond well to a lower-dose intervention. Success with integrating Fitbit MVPA data into the electronic health record (EHR) with the capability to provide weekly progress feedback to participants via the EHR's patient portal represents a relatively low resource (vs. coaching or supervised exercise) and potentially efficacious minimal intervention that could be augmented as needed. Placement of the intervention within the EHR is a major advance because it communicates that MVPA is central to survivors' health and is a priority of the cancer care team. Clinicians can be engaged to ensure the intervention is viewed as integral to survivorship care with minimal burden by referring patients to an EHR-based intervention, endorsing intervention messages delivered via the EHR and reviewing a patient's progress at their clinic visits using simple EHR alerts.

While the Fitbit plus EHR integration (Fitbit+EHR) minimal intervention will be sufficient for some survivors to increase their MVPA, others will need more support. Little data exists to determine what strategies would be most effective for augmenting a minimal intervention. Further, it is unknown how long the minimal intervention should be continued before augmentations are used. Some survivors may need more support early on, while others may initially succeed but later fail as the weekly MVPA goal increases. Still others may falter initially and recover.

This project uses an innovative adaptive experimental approach, to determine the optimal augmentation tactics to the minimal (Fitbit+EHR) MVPA intervention in inactive breast and endometrial cancer survivors (n=320). All women will receive the Fitbit+EHR intervention. Those who do not respond (meet ≤80% of MVPA goal over previous 4 weeks) will be randomized to one of two more intensive augmentation tactics using technology, alone, or in combination with a more traditional component: (1) online gym with access to exercise videos or (2) coaching calls. Participants in the minimal intervention will be evaluated for non-response every 4 weeks so augmentation is delivered when they lapse. Responders will continue with the minimal intervention. The primary outcome is accelerometer-measured weekly minutes of MVPA at 6 months, 12 months, and 30 months. The investigator will also examine the effects of the intervention sequences on symptom burden and functional performance, important indicators of morbidity in these populations.

This is the first systematic effort to develop an adaptive MVPA intervention in any cancer population. Knowledge gained from this study will inform the development of effective, scalable clinic-based interventions to improve quality of life and reduce disease burden among breast and endometrial cancer survivors.

[Protocol Amendment approved on 5/24/2023 added a 30 month time point to data collection.]

ELIGIBILITY:
Inclusion Criteria:

* Female adult (≥18 years of age)
* Diagnosis of Stage I-III breast or Stage I-II Type 1 endometrial cancer within the past 5 years.
* At least 3 months past completion of primary active treatment (i.e., surgery, chemotherapy, and/or radiation). May still be undergoing endocrine or Human epidermal growth factor receptor 2 (Her2) therapies.
* Insufficiently active, defined as ≤60 min/week of MVPA, performed in bouts of ≥10 minutes.This is 40% of the recommended amount of MVPA based on the 2008 Federal Guidelines and the American Cancer Society's guidelines for cancer survivors. The 7-Day Recall will be used to screen for physical activity; eligibility will be confirmed prior to randomization using the ActiGraph accelerometer.
* Able to access high-speed Internet daily at home on a computer, smartphone, or tablet. Internet access may be through a household connection or a wireless provider (e.g., Verizon, AT&T). For compatibility with the Fitbit, the device must run a Windows, Apple, or Android operating system.
* Have a MyChart account or be willing to create one.
* Fluent in spoken and written English language.
* For safety, participants will be screened using the Physical Activity Readiness Questionnaire (PAR-Q) and the Falls Risk Screener, which address joint and cardiovascular problems, balance issues, and other concerns. Physician consent will be obtained for all participants who meet the following criteria:

  * Answer yes to ≥1 question on the PAR-Q OR
  * Answer yes to ≥4 questions on the Falls Risk Screener
* Willing and able to attend study visits at the University of Wisconsin, Madison or Northwestern University, Chicago
* Own and can use a smartphone

Exclusion Criteria:

* Any absolute contraindications to exercise (i.e. acute myocardial infarction, severe orthopedic conditions), metastatic disease or planned elective surgery during intervention/ follow-up.
* Self-reported difficulty transitioning walking 1 block (as a proxy measure of basic physical functioning), or inability to work towards the intervention goals
* Plans to become pregnant or to move from the area within the next two years
* Current enrollment in another dietary or physical activity trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 323 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change in the 'Weekly minutes of moderate- to-vigorous physical activity (MVPA)' as measured by actigraph | Baseline, 6 months, 12 months, 30 months
  Change in the 'Weekly minutes of moderate- to-vigorous physical activity (MVPA)' as measured by actigraph
Change in the 'Weekly minutes of MVPA' as measured by Fitbit | Baseline, 6 months, 12 months, 30 months
  Change in the 'Weekly minutes of moderate- to-vigorous physical activity (MVPA)' as measured by Fitbit
Change in the 'Weekly minutes of MVPA' as reported in Self-report | Baseline, 6 months, 12 months, 30 months
  Change in the 'Weekly minutes of moderate- to-vigorous physical activity (MVPA)' as reported in Self-report
Godin Leisure Time Exercise Questionnaire (GLTEQ) score | 12 months and 30 months
  Godin Leisure Time Exercise Questionnaire (GLTEQ) score measures the number of times on average a person does strenuous/moderate/mild exercise for more than 15 minutes during their leisure time.
  Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light)
  GLTEQ Score Interpretation 24 units or more - Active 14 - 23 units - Moderately Active Less than 14 units - Insufficiently Active/Sedentary
Change in the 'Sitting time per week' | Baseline, 6 month, 12 month, 30 months
  Although not a measure of physical activity, the Sitting Time Questionnaire will be administered at each of the three main data collection time points to provide context for the participant's inactive time.
  Less sitting time per week correlates to more physical activity

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPB) score | Baseline, 6 months, 12 months, 30 months
  Participants will complete the Short Physical Performance Battery (SPB), a well-validated physical function performance measure. This battery assesses lower extremity function in adults.
  The SPB score is based on timed measures of gait speed, ability to rise from a chair, and standing balance. Gait speed will be measured using the better of two recorded times over a 4-meter course. Chair stand time will be measured as the time needed to rise five times from a seated position in a chair, with arms folded across the chest. For the balance test, participants will be asked to maintain their feet side-by-side, semi-tandem, and tandem positions for 10 seconds each. Each individual performance measure will be scored according to established cutpoints and aggregated for a total SPB score.
  Total SPB score range: 0 (worst performance) to 12 (best performance).
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) short form score for physical function | Baseline, 6 months, 12 months, 30 months
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life that are known to be common long-lasting symptoms after cancer treatment.
  At each time point, participants will complete PROMIS short form measures for physical function.The functional performance tests are in-person tests that assess physical abilities (strength, mobility) in ways that are relevant to daily living. PROMIS measures are measured on T-score metrics.
  The short form consists of 20 questions which can be answered on a scale of 1-5 where 1-Unable to do, 2-with much difficulty, 3-with some difficulty,4-with a little difficulty, 5- without any difficulty. The cumulative score ranges from 20 to 100, where higher scores correlates to more physically active person.
Change in PROMIS short form score for fatigue | Baseline, 6 months, 12 months, 30 months
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life that are known to be common long-lasting symptoms after cancer treatment. The functional performance tests are in-person tests that assess physical abilities in ways that are relevant to daily living.
  Fatigue short form has 8 items. Each item on the measure is rated on a 5-point scale( 1-Not at all, 2-A little bit, 3-Somewhat, 4-Quite a bit, 5-Very much) with a range in score from 8 to 40 with higher scores indicating more fatigue
Change in PROMIS short form score on Sleep Related Impairment | Baseline, 6 months, 12 months, 30 months
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life that are known to be common long-lasting symptoms after cancer treatment. The functional performance tests are in-person tests that assess physical abilities in ways that are relevant to daily living.
  Sleep related impairment short form has 8 items. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater sleep disturbance.
Change in PROMIS short form score on Sleep Disturbance | Baseline, 6 months, 12 months, 30 months
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life that are known to be common long-lasting symptoms after cancer treatment. The functional performance tests are in-person tests that assess physical abilities in ways that are relevant to daily living.
  PROMIS sleep disturbance short form has 8 items. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Change in PROMIS short form score on Applied Cognition-Abilities | Baseline, 6 months, 12 months, 30 months
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life that are known to be common long-lasting symptoms after cancer treatment. The functional performance tests are in-person tests that assess physical abilities in ways that are relevant to daily living.
  Applied Cognition-Abilities short form has 8 items. Each item on the measure is rated on a 5-point scale (1-Very much; 2-Quite a bit; 3-Somewhat; 4-A little bit, 5-Not at all) with a range in score from 8 to 40. Higher score correlates to higher cognitive ability
Change in PROMIS short form score for Emotional Distress - Anxiety | Baseline, 6 months, 12 months, 30 months
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life that are known to be common long-lasting symptoms after cancer treatment. The functional performance tests are in-person tests that assess physical abilities in ways that are relevant to daily living.
  Emotional Distress- Anxiety has 7 items. Each item on the measure is rated on a 5-point scale (1-never; 2-rarely; 3-sometimes. 4-often; 5-always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
Change in PROMIS short form score for Depression | Baseline, 6 months, 12 months, 30 months
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life that are known to be common long-lasting symptoms after cancer treatment. The functional performance tests are in-person tests that assess physical abilities in ways that are relevant to daily living.
  PROMIS short form for Depression has 8 items. Each item on the measure is rated on a 5-point scale (1-never, 2-rarely, 3-sometimes; 4-often, 5-always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Change in PROMIS short form score for Emotional Support | Baseline, 6 months, 12 months, 30 months
  PROMIS Emotional Support scale is an 8-item scale. Individual items are scored from 1-5. The total range of possible overall raw scores is 8-40. These are then translated to T-scores using a table provided by PROMIS. The possible range of T-scores is 24.7-63.5. Emotional support may predict the adherence to the intervention.
Change in FACT-B Quality of Life Survey | Baseline, 6 months, 12 months, 30 months
  The Functional Assessment of Cancer Therapy - Breast (FACT-B) Quality of Life Survey is a 37-item survey scored on a 5-point likert scale where 0 is 'not at all' to 4 is 'very much'. The total possible range of scores is 0-148 where lower scores indicate improved quality of life.
Change in FACT-En Quality of Life Survey | Baseline, 6 months, 12 months, 30 months
  The Functional Assessment of Cancer Therapy - Endometrial (FACT-En) Quality of Life Survey is a 43-item survey scored on a 5-point likert scale where 0 is 'not at all' to 4 is 'very much'. The total possible range of scores is 0-172 where lower scores indicate improved quality of life.

OTHER OUTCOMES:
Social Cognitive Theory (SCT) constructs : Exercise Self-Efficacy Scale | 12 months
  Self-efficacy will be assessed using the Exercise Self-Efficacy Scale which assess the beliefs of participants to be able to exercise in the future.
  Scale consists of 6 questions which are graded from 0-100% in gradation of 10. 0% correlates to 'not at all confident' whereas 100% means highly confident in continuing their exercise.
SCT constructs : Barriers specific Self-Efficacy scale | 12 months
  Self-efficacy will be assessed using the Barriers Self-Efficacy Scale which assess the beliefs in ability to be active over the next 12 weeks, despite common barriers.
  Items in the scale reflect situations which can be common reasons for preventing participants from actively exercising or, in some cases, dropping out. Scale has 13 questions which are graded from 0-100% in gradation of 10. 0% correlates to 'not at all confident' whereas 100% means Highly confident in continuing their exercise in the situations listed in the questionnaire. Scores can range from 0-1300 where higher scores means more adherence to the exercise regime in the event of unfavorable conditions.
SCT constructs : Physical activity enjoyment scale | 12 months
  Physical Activity Enjoyment Scale which assesses level of enjoyment and satisfaction with current MVPA program will be used to measure facilitators/barriers.
  The scale consists of 18 questions which can be answered on a scale of 1-7(I enjoy it- I hate it). The cumulative score ranges from 18-126 where higher scores means participant is not enjoying the physical activity.
SCT constructs : Exercise goal setting scale | 12 months
  The Exercise Goal Setting Scale will assess MVPA-related exercise goal-setting. Questionnaire contains 10 questions which can be answered in the grading of 'Does not describe'/ 'Describe moderately'/ 'Describe completely'. Based on the response score on the exercise goal setting scale can range from 10-50. Higher scores correlates to firmer exercise goals.
Social Cognitive Theory (SCT) constructs :Multidimensional Outcome Expectations for Exercise Scale(MOESS) | 12 months
  MOESS is used to assess three related, but conceptually independent domains of outcome expectations for exercise (i.e., physical, social, and self-evaluative outcome expectations). For each item, participants indicate the degree to which they agree with each statement.
  The scale consists of 20 questions which can be answered as 1-Strongly agree, 2-Disagree, 3-Neutral, 4-Agree, 5-Strongly agree. Higher scores correlates to higher outcome expectation for exercise.
Social Cognitive Theory (SCT) constructs : Social Support for Exercise Scale | 12 months
  The Social Support for Exercise Scale which assesses support for MVPA received from friends, family and other survivors.
  Scale contains 10 questions which can be answered as:1-Never, 2-Rarely, 3-A few times, 4-Often, 5-Very Often, 8-Does not apply.
  Scale includes separate categories for support by Family, Friends and Other survivors. Applicable scores can range from 10-50. Higher scores(max 50 in the applicable range) in each category correlates to stronger social support for exercise from that group.
Intervention implementation and fidelity: Fitbit wear time per week | up to 12 months
  Intervention implementation and fidelity: Fitbit wear time per week
Intervention implementation and fidelity: number of read/unread emails | up to 6 months
  Status of feedback emails delivered via the EHR's patient portal will be measures as number of read/unread emails
Intervention implementation and fidelity: Number of feedback emails delivered via the EHR's patient portal | up to 12 months
  Intervention implementation and fidelity: Number of feedback emails delivered via the EHR's patient portal
Intervention implementation and fidelity: Time spent in watching online gym exercise videos | up to 12 months
  Intervention implementation and fidelity: Time spent in watching online gym exercise videos
HINTS Questionnaire | Baseline, 6 months, 12 months
  The Health Information National Trends Survey (HINTS) will be used in part to measure the intervention implementation and fidelity. HINTS collects nationally representative data routinely about the American public's use of cancer-related information. It is a 30-item multiple choice survey about medical research and medical records and patient-provider communications.
Participant Program Evaluation | up to 12 months
  The participant program evaluation is designed to get feedback from participants. It contains multiple different question types across 16-items about the intervention, and 7-items about the coaching calls, and 17-items about the online gym experience.
Clinician Questionnaire | Baseline, 6 months, 12 months (and every 6 months thereafter until data collection is complete)
  The clinician questionnaire surveys clinicians about their experience with the intervention. This questionnaire contains a variety of questions on different 5 point likert scales as well as open ended queries for feedback on the intervention.
Change in Virtual Functional Performance Testing Feedback Survey | Baseline, 6 months, 12 months
  The Virtual Functional Performance Testing Feedback Survey includes a mixture of multiple choice and free response (6 items), and 5 point likert items (15 items). It is intended as a feedback measure from participants in response to the virtual aspects of this intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Pickett, Ph.D., Principal Investigator — University of Wisconsin, Madison; Siobhan Phillips, Ph.D., MPH, Principal Investigator — Northwestern University, Chicago
Locations (2):
- United States (2):
  - Department of Preventative Medicine, Northwestern University, Chicago, Illinois
  - Department of Kinesiology, University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cadmus-Bertram L, Solk P, Agnew M, Starikovsky J, Schmidt C, Morelli WA, Hodgson V, Freeman H, Muller L, Mishory A, Naxi S, Carden L, Tevaarwerk AJ, Wolter M, Barber E, Spencer R, Sesto ME, Gradishar W, Gangnon R, Spring B, Nahum-Shani I, Phillips SM. A multi-site trial of an electronic health integrated physical activity promotion intervention in breast and endometrial cancers survivors: MyActivity study protocol. Contemp Clin Trials. 2023 Jul;130:107187. doi: 10.1016/j.cct.2023.107187. Epub 2023 Apr 21. PMID 37086916